CLINICAL TRIAL: NCT05223881
Title: 13^C-Spirulina Platensis Gastric Emptying Breath Test for Diagnosis of Gastroparesis in Patients With Cystic Fibrosis
Brief Title: Gastroparesis in Cystic Fibrosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is not feasible at this time due to staffing limitations
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Daphna Katz, Pediatric Gastroenterology Fellow, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20211043
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Gastroparesis
Keywords: Cystic Fibrosis; Pediatrics; Altered lung function
MeSH Terms: conditions — Gastroparesis; Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cystic Fibrosis (Experimental): Patients who are diagnosed with Cystic Fibrosis.
  Interventions: Device: 13^C Spirulina Platensis Gastric Emptying Breath Test (GEBT)
- Healthy Normal (Active Comparator): Patients in this arm will be a sibling of patients who have been diagnosed with Cystic Fibrosis.
  Interventions: Device: 13^C Spirulina Platensis Gastric Emptying Breath Test (GEBT)

INTERVENTIONS:
Device: 13^C Spirulina Platensis Gastric Emptying Breath Test (GEBT) — After an overnight (minimum 8 hours) fast, patients are given a standardized test meal, after which they are administered the GEBT. Patients are asked to hold a glass tube in a comfortable position, take a deep breath and pause momentarily, blow gently into the tube for 5 - 10 seconds, slowly withdraw straw from tube while continuing to breath into tube, and immediately close the tube securely with the cap.

SUMMARY:
The purpose of this research is to determine if an investigational device called the 13C-Spirulina Gastric Emptying Breath Test (GEBT), can accurately diagnose gastroparesis (delayed emptying of the stomach) in patients with Cystic Fibrosis (CF).

ELIGIBILITY:
Inclusion Criteria:

* Patients age 4 years* and above with a genetically confirmed diagnosis of CF (*This age was chosen as patients younger than 4 years rarely undergo GES)
* Actively being followed at the University of Miami CF Center (i.e. seen within the past 5 years at a University of Miami pediatric or adult pulmonology clinic)

Exclusion Criteria:

* History of abdominal surgeries involving gastrointestinal luminal resection (i.e. small bowel or colonic resection that increases risk of post-operative strictures or narrowing of the lumen). Nissen fundoplication, gastrostomy tube placement, gynecologic surgeries, appendectomy, and/or cholecystectomy are not excluded.
* Gastrointestinal comorbidities that impact absorption such as Inflammatory Bowel Disease and Celiac Disease
* Known hypersensitivity to Spirulina, egg, milk or wheat allergens
* Patients not able to consume at least 50% of a standard test meal
* Pregnant women
* Adults unable to consent
* Prisoners

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-14 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Rate of gastric emptying | 4 hours
  The kPCD value (13CO2 excretion rate) at any time t, is proportional to the rate of gastric emptying. Increasing kPCD values represent increasing rates of gastric emptying.

SECONDARY OUTCOMES:
Rate of gastric emptying over time | 6 months
  The kPCD value (13CO2 excretion rate) at any time t, is proportional to the rate of gastric emptying. Increasing kPCD values represent increasing rates of gastric emptying.

CONTACTS AND LOCATIONS:
Overall Officials: Daphna Katz, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No